CLINICAL TRIAL: NCT00599118
Title: Identification of Genetic, Biochemical and Hormonal Factors Contributing to Atrial Fibrillation
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mina Chung, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 8271
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Genetics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, buffy coat, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- atrial fibrillation: Atrial fibrillation
- Control: Control subjects with no atrial fibrillation

SUMMARY:
The purpose of this study is to establish a genebank repository of blood samples and data to generate information about the hereditary (genetic) basis of atrial fibrillation.

DETAILED DESCRIPTION:
Blood samples and data will be collected from subjects with atrial fibrillation and normal controls. The primary aim of future research using these samples is to identify mechanisms and pathogenesis of atrial fibrillation. Through this information, we hope to identify targets for new therapies and improve knowledge and understanding of atrial fibrillation. Identification of disease genes could improve strategies that prevent progression of atrial fibrillation to more persistent disease.

ELIGIBILITY:
Inclusion Criteria for Atrial Fibrillation group:

* Male or female at least 18 years old
* Subjects with a history of or current Atrial Fibrillation
* Subjects able to give informed consent Exclusion Criteria for Atrial Fibrillation group: no history of atrial fibrillation

Inclusion Criteria for Controls:

* Male or female at least 18 years old
* Subjects with no history of Atrial Fibrillation
* Subjects able to give informed consent Exclusion Criteria for controls: History of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants associated with atrial fibrillation | Baseline
  Genome-wide association study of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Mina K Chung, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinical Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No